CLINICAL TRIAL: NCT00838175
Title: Characteristics Predictive of Success and Complications in the Use of Suture-Mediated Closure of Femoral Venous Access
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Andrew C. Eisenhauer, MD, Brigham and Women's Hospital
Other Study IDs: 2007P-001023
Record Dates: First submitted 2009-02-04; First posted 2009-02-06 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Cardiac Catheterization
Keywords: Peripheral Venous Catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All pts. who have undergone percutaneous intervention who received a suture-mediated closure of the venous access site will be screened for eligibility for this research trial.
  Interventions: Procedure: suture mediated closure

INTERVENTIONS:
Procedure: suture mediated closure — Suture mediated closure of femoral venous access
  Other Names: Suture mediated closure of femoral venous access

SUMMARY:
Suture-mediated closure devices are effective and safe for achieving rapid hemostasis in femoral venous access site and reducing the incidence of complications associated with traditional closure methods. Furthermore, there are predictive factors(such as sheath size, obesity, procedure duration, and anticoagulation status)that we can use to assess the procedure's likelihood of success in various patients.

DETAILED DESCRIPTION:
This is a retrospective cohort study of consecutive patients receiving suture-mediated closure of the femoral vein following catheterization. All patients undergoing cardiac or arterial catheterization by the Interventional Cardiovascular Medicine Service at The Brigham and Women's hospital from 3/1/02 to the onset of the study and who had femoral venous access during that time were considered for closure of the venous site; however, the decision to use the closure device was left to the discretion of the physician. Contraindications to using the closure device include a groin hematoma that had developed during the procedure and/or difficult access due to extensive scar tissue from surgery or multiple prior vascular accesses.

All in-hospital endpoints have been collected in the pre-existing Catheterization Laboratory Database. Patient's data will be extracted from this database as indicated in the procedure below. Each patient will be reviewed for clinical follow-up and the presence of adverse events including but not limited to hematoma, thrombosis, blood loss, vascular imaging, the need for additional procedures, and re-admissions within 30 days of closure. If necessary, further data will be collected via a phone interview with the patients. Univariate and multivariate analysis will be performed to determine the factors that predict inadequate or incomplete closure or the development of complications mentioned in the section above. A predictive model based on the identified risk factor will be developed and tested prospectively in the next phase of this ongoing investigation.

ELIGIBILITY:
Inclusion Criteria:

* All consented pts. over the age of 18 who received sutured mediated femoral vein following catheterization

Exclusion Criteria:

* Pt.s who are unable to give consent.
* Pts. whose participation in research is contraindicated for medical reasons are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult over the age of 18, who received a suture mediated closure of the femoral vein following catheterizaton at the BWH cath lab.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-02 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
To determine the safety and effectiveness of the suture-mediated closure devices in closing femoral venous access sites. | Within 30 days of procedure/closure

SECONDARY OUTCOMES:
To identify factors that are predictive of success and failure of the suture mediated closures. | Within 30 days of procedure/closure

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C Eisenhauer, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States